CLINICAL TRIAL: NCT02461719
Title: Multicenter, Randomized, Double-blind phⅢ Study of TJCS Eye Drops Group and Restasis Eye Drops Group for 12 Weeks After Treatment, Each Treatment Group Comparisons for Evaluation of Efficacy and Safety in Moderate to Severe Dry Eye Disease.
Brief Title: Efficacy and Safety Study of TJCS for Treatment of Moderate to Severe Dry Eye Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJCS_P3
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYPORIN N EYE DROPS 0.05%(TJCS eye drop) (Experimental): CYPORIN N EYE DROPS 0.05%(TJCS eye drop) 1 drop twice/day for 12 weeks to both eyes
  Interventions: Drug: CYPORIN N EYE DROPS 0.05%(TJCS eye drop)
- Restasis eye drop (Active Comparator): Restasis eye drop(Cyclosporine ophthalmic solution 0.05%) 1 drop twice/day for 12 weeks to both eyes
  Interventions: Drug: Restasis

INTERVENTIONS:
Drug: CYPORIN N EYE DROPS 0.05%(TJCS eye drop) — 1 drop twice/day for 12 weeks to both eyes.
  Other Names: Cyclosporine Eye Drops(CYPORIN N)
  Arms: CYPORIN N EYE DROPS 0.05%(TJCS eye drop)
Drug: Restasis — 1 drop twice/day for 12 weeks to both eyes. Invert the unit dose vial a few times to obtain a uniform, white, opaque emulsion before using.
  Other Names: Cyclosporine Eye Drops (Restasis)
  Arms: Restasis eye drop

SUMMARY:
The purpose of this clinical Study is TJCS Eye Drops 0.05%(Cyclosporine ophthalmic nano-emulsion) group and Restasis Eye Drops 0.05%(Cyclosporine ophthalmic suspension) group 12 weeks after treatment, each treatment group comparisons for evaluation of efficacy and safety in Moderate to Severe Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Patients with moderate to severe dry eye
* Screening both eyes, the corrected visual acuity is 0.2 or more

Exclusion Criteria:

* Screening visits within 4 weeks who treated with systemic cyclosporine or topical cyclosporine ophthalmic solutions.
* Screening visits within 2 months the patients with systemic or ocular disorders affected the test results (ocular surgery, trauma, or disease)
* Intraocular pressure(IOP)> 25 mmHg
* Patient using or to use punctual plug within 1 months.
* Patients with contact lens.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Corneal staining test | 12 weeks

SECONDARY OUTCOMES:
Corneal staining test | 4, 8 weeks
Conjunctival staining | 4, 8, 12 weeks
Corneal and Conjunctival staining sum Score | 4, 8, 12 weeks
Ocular surface disease index (OSDI) | 4, 8, 12 weeks
Tear break up time (TBUT) | 4, 8, 12 weeks
Non-anesthetic Schirmer test | 4, 8, 12 weeks
Frequency of concurrent drug use | 4, 8, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, South Korea